CLINICAL TRIAL: NCT00005811
Title: A Phase II Study of Intrathecal Topotecan (NSC #609699) in Patients With Refractory Meningeal Malignancies
Brief Title: Topotecan Hydrochloride in Treating Children With Meningeal Cancer That Has Not Responded to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01848; P9962; U10CA098543 (NIH); CDR0000067813 (Registry Identifier: PDQ (Physician Data Query)); NCT00013676 (obsolete NCT alias)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Diffuse Mixed Cell Lymphoma; AIDS-related Diffuse Small Cleaved Cell Lymphoma; AIDS-related Immunoblastic Large Cell Lymphoma; AIDS-related Lymphoblastic Lymphoma; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; AIDS-related Small Noncleaved Cell Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; HIV-associated Hodgkin Lymphoma; Leptomeningeal Metastases; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Meningeal Carcinomatosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Burkitt Lymphoma; Recurrence | interventions — Topotecan; trioctyl phosphine oxide

ARMS (1):
- Treatment (topotecan hydrochloride) (Experimental): INDUCTION: Patients receive topotecan hydrochloride IT over 5 minutes twice weekly for 6 weeks.
  CONSOLIDATION: Beginning 1 week after completion of induction, patients receive topotecan hydrochloride IT over 5 minutes weekly for 4 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Beginning 2 weeks after completion of consolidation, patients receive topotecan hydrochloride IT over 5 minutes twice monthly for 4 months and then monthly through year 1.
  Interventions: Drug: topotecan hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: topotecan hydrochloride — Given IT
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. This phase II trial is studying how well topotecan hydrochloride works in treating children with meningeal cancer that has not responded to previous treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the therapeutic activity of intrathecal topotecan, in terms of response rate and time to central nervous system (CNS) progression, in pediatric patients with recurrent or refractory neoplastic meningitis.

II. Determine the safety and toxicity of this regimen in these patients. III. Evaluate the concentration of matrix metalloproteinases (MMPs) in the cerebrospinal fluid (CSF) of these patients.

OUTLINE: Patients are stratified according to disease type (acute lymphoblastic leukemia vs. other leukemia/lymphoma vs medulloblastoma vs other solid tumors). (Recurrent CNS acute lymphoblastic leukemia stratum only open to accrual as of 11/30/04)

INDUCTION: Patients receive topotecan hydrochloride intrathecally (IT) over 5 minutes twice weekly for 6 weeks.

CONSOLIDATION: Beginning 1 week after completion of induction, patients receive topotecan hydrochloride IT over 5 minutes weekly for 4 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Beginning 2 weeks after completion of consolidation, patients receive topotecan hydrochloride IT over 5 minutes twice monthly for 4 months and then monthly through year 1.

After completion of study treatment, patients are followed up monthly for 3 months, every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 14-77 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven refractory leukemia, lymphoma, or other solid tumor thathas overt meningeal involvement (Recurrent CNS acute lymphoblastic leukemia stratum only open to accrual as of 11/30/04)

  * Definition of meningeal disease:

    * Leukemia/lymphoma (including acute lymphoblastic leukemia)

      * CSF cell count greater than 5/mm^3 AND evidence of blast cells oncytospin preparation or by cytology
      * Refractory to conventional therapy, including radiotherapy (i.e., in second or greater relapse)
      * No concurrent bone marrow relapse
    * Solid tumors (including medulloblastoma)

      * Presence of tumor cells on cytospin preparation or cytology OR presence ofmeningeal disease on MRI scans
* No clinical evidence of obstructive hydrocephalus or compartmentalization ofCSF flow as documented by radioisotope indium In 111 or technetium Tc 99 DTPAflow study

  * If CSF flow block is demonstrated, focal radiotherapy must be administered tosite of block to restore flow and a repeat CSF flow study must show clearing of blockage
* No ventriculoperitoneal or ventriculoatrial shunt unless:

  * Patient is shunt independent and there is evidence that the shunt is nonfunctional
  * CSF flow study demonstrates normal flow
* No impending cord compression, CNS involvement requiring local radiotherapy(e.g., optic nerve), or isolated bulky ventricular or leptomeningeal basedlesions
* Performance status - Lansky 50-100% (age 10 and under)
* Performance status - Karnofsky 50-100% (over age 10)
* At least 8 weeks
* Platelet count greater than 40,000/mm^3 (transfusions allowed)
* Bilirubin less than 2.0 mg/dL
* SGPT less than 5 times normal
* Creatinine less than 1.5 mg/dL
* Electrolytes, calcium, and phosphorus normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant illness (e.g., uncontrolled infection, except HIV [i.e., AIDS-related lymphomatous meningitis])
* Prior immunotherapy allowed and recovered
* At least 3 weeks since systemic CNS directed chemotherapy (6 weeks for nitrosoureas) and recovered
* At least 1 week since prior intrathecal (IT) chemotherapy (2 weeks for cytarabine [liposomal])
* No prior IT chemotherapy on days -14 to -7 before study entry unless evidence of disease progression (e.g., increasing WBC and percentage blasts in patients with leukemia/lymphoma or increased leptomeningeal enhancements in patients with solid tumors) (Recurrent CNS acute lymphoblastic leukemia stratum only open to accrual as of 11/30/04)
* Concurrent chemotherapy to control systemic disease or bulk CNS disease allowed if the systemic chemotherapy is not a phase I study agent that significantly penetrates the CSF (e.g., high-dose systemic methotrexate [greater than 1 g/m^2], thiotepa, high-dose cytarabine, temozolomide, IV mercaptopurine, nitrosourea, or topotecan) or an agent known to have serious unpredictable CNS side effects
* Concurrent dexamethasone or prednisone allowed if part of a systemic chemotherapy regimen
* See Disease Characteristics
* At least 8 weeks since prior cranial irradiation and recovered
* No concurrent whole brain or craniospinal irradiation
* At least 7 days since prior investigational drug

  * Time period should be extended if patient has received any investigational agent that is known to have delayed toxic effects after 7 days or a prolonged half-life
* No other concurrent investigational agents
* No concurrent therapy (IT or systemic) for leptomeningeal disease
* No other concurrent systemic agents that significantly penetrate the blood-brain barrier

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2000-04; Primary Completion 2006-04 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
For the leukemia and lymphoma patients, an objective response rate, defined to be the proportion of Complete Responses of less than 0.10 | Up to 54 months
For the patients with solid tumors, a proportion of patients who do not experience an event, defined to be death, progressive disease, relapse, or second malignancy of less than 0.3 | Up to 54 months
Safety and toxicity | Up to 54 months
Concentration of matrix metalloproteinases in the CSF | Up to 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States